CLINICAL TRIAL: NCT05723835
Title: A Study Evaluating the Safety and Efficacy of Once-weekly Dosing of Somapacitan in a Basket Study Design in Paediatric Participants With Short Stature Either Born Small for Gestational Age or With Turner Syndrome, Noonan Syndrome or Idiopathic Short Stature
Brief Title: A Research Study Looking at How Safe Somapacitan is and How Well it Works in Children Who Need Help to Grow - REAL 9
Acronym: REAL 9
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4469; U1111-1277-9765 (Other: World Health Organization (WHO)); 2022-501055-87 (EudraCT Number)
Record Dates: First submitted 2023-01-29; First posted 2023-02-13 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: SGA; Turner Syndrome; Noonan Syndrome; ISS
MeSH Terms: conditions — Turner Syndrome; Noonan Syndrome | interventions — somapacitan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Somapacitan (Experimental): Participants will receive Somapacitan for 26-week main phase followed by 130-week extension phase.
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — Somapacitan 0.24 milligrams per kilograms per week (mg/kg/week) will be administered subcutaneously (s.c.) using PDS290 pen-injector.

SUMMARY:
The purpose of this study is to find out if somapacitan is safe and how well somapacitan works in children either born small for gestational age or with Turner syndrome, Noonan syndrome or idiopathic short stature. Somapacitan is a new growth hormone medicine for treatment of low level of growth hormone. The study will last for about 3 years. During the study, the participants will be treated with somapacitan once a week. Somapacitan can be injected anytime during the day. The study doctor or nurse will show how to inject somapacitan, so that the participant knows how to do it at home.

ELIGIBILITY:
Inclusion Criteria:

Applicable to children with SGA:

* Born small for gestational age (birth length below -2 SDS OR birth weight below -2 SDS OR both) (according to national standards).
* Age:

  - Male participants: Age equal to or above 11.0 years and below 18.0 years at screening.

  - Female participants: Age equal to or above 10.0 years and below 18.0 years at screening.
* Open epiphyses; defined as bone age less than (<) 14 years for females and bone age < 16 years for males.
* For Growth Hormone (GH) treatment naïve participants: Impaired height defined as at least 2.5 standard deviations below the mean height for chronological age and sex at screening according to the standards of Centers for Disease Control and Prevention.

Applicable to children with TS:

• Diagnosis of TS according to local clinical practice.

* Age:

  - Female participants: Age equal to or above 10.0 years and below 18.0 years at screening.
* Open epiphyses; defined as bone age < 14 years for females and bone age < 16 years for males.
* For GH treatment naïve participants: Impaired height defined as at least 2.0 standard deviation below the mean height for chronological age and sex at screening according to the standards of Centers for Disease Control and Prevention.
* For GH treatment naïve participants: Confirmed diagnosis of TS by 30-cell (or more) lymphocyte chromosomal analysis or confirmation of TS and TS mosaicism using comparative genomic hybridization (CGH)-array.

Applicable to children with NS:

* Diagnosis of NS according to local clinical practice.
* Age:

  * Male participants: Age equal to or above 11.0 years and below 18.0 years at screening.
  * Female participants: Age equal to or above 10.0 years and below 18.0 years at screening.
* Open epiphyses; defined as bone age < 14 years for females and bone age < 16 years for males.
* For GH treatment naïve participants: Clinical diagnosis of NS according to van der Burgt score list and genetic test result or confirmed mutation in any of the genes associated with NS before allocation.

Applicable to children with ISS:

* Age:

  - Male participants: Age equal to or above 11.0 years and below 18.0 years at screening.

  - Female participants: Age equal to or above 10.0 years and below 18.0 years at screening.
* Open epiphyses; defined as bone age < 14 years for females and bone age < 16 years for males.
* For GH treatment naïve participants: Impaired height defined as at least 2.5 standard deviations below the mean height for chronological age and sex at screening
* For GH treatment naïve participants: Normal GH secretion (GH peak above 7 ng/mL) during GH stimulation test performed within 18 months prior to screening.
* For GH treatment naïve participants: Bone age not delayed more than 2 years compared to chronological age at screening.

Exclusion Criteria:

* Children with suspected or confirmed growth hormone deficiency according to local practice.
* Children diagnosed with diabetes mellitus or screening values from the central laboratory.
* Fasting plasma glucose above or equal to 126 milligrams per deciliter (mg/dL) [7.0 millimoles per litre (mmol/L)] or
* Glycated hemoglobin (HbA1c) above or equal to 6.5%.
* Current inflammatory diseases requiring systemic corticosteroid treatment for longer than 2 consecutive weeks within the last 3 months prior to screening.
* Children requiring inhaled glucocorticoid therapy at a dose greater than 400 micrograms per day (µg/day) of inhaled budesonide or equivalent (i.e., 250 µg/day for fluticasone propionate) for longer than 4 consecutive weeks within the last 12 months prior to screening.
* History or known presence of malignancy including intracranial tumours.

Applicable to children with SGA:

• Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with height, such as, but not limited to:

* Poorly controlled or uncontrolled hormonal deficiencies.
* Known chromosomal aneuploidy or significant gene mutations causing medical 'syndromes' with short stature, including but not limited to Laron syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, skeletal dysplasias, abnormal short stature homeobox (SHOX) gene analysis or absence of GH receptors.

Applicable to children with TS:

• Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with height, such as, but not limited to:

* Known family history of skeletal dysplasia.
* Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants.
* Any other disorder that can cause short stature such as, but not limited to nutritional disorders, chronic systemic illness and chronic renal disease.
* Mosaicism below 10%.
* TS with Y-chromosome mosaicism where gonadectomy has not been performed.
* New York Heart Association (NYHA) class II or above or requiring medication for any heart condition.

Applicable to children with NS:

• Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with height, such as, but not limited to:

* Known family history of skeletal dysplasia.
* Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants.
* Any other disorder that can cause short stature such as, but not limited to nutritional disorders, chronic systemic illness and chronic renal disease.
* Noonan-related disorders including but not limited to: Noonan syndrome with multiple lentigines (formerly called 'LEOPARD' syndrome), Noonan syndrome with loose anagen hair, cardiofaciocutaneous syndrome (CFC), Costello syndrome, neurofibromatosis type 1 (NF1) and Legius syndrome.

Applicable to children with ISS:

• Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with height, such as, but not limited to:

* Known family history of skeletal dysplasia.
* Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants.
* Any other disorder that can cause short stature such as, but not limited to nutritional disorders, chronic systemic illness and chronic renal disease.
* Poorly controlled or uncontrolled hormonal deficiencies.
* Known chromosomal aneuploidy or significant gene mutations causing medical 'syndromes' with short stature, including but not limited to Laron syndrome, Prader-Willi syndrome, Russell-Silver Syndrome, skeletal dysplasias, abnormal SHOX gene analysis or absence of GH receptors.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2027-10-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (17):
- United States (6):
  - Univ of AL at Birmingham_BRM, Birmingham, Alabama
  - Sutter Valley Med Fdt Ped Endo, Sacramento, California
  - Rocky Mt Ped and Endo, Centennial, Colorado
  - Childrens National Medical Ctr, Washington D.C., District of Columbia
  - Rocky Mt Clin Res, LLC, Idaho Falls, Idaho
  - Children's Minnesota, Saint Paul, Minnesota
- Malaysia (2):
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - University Technology MARA (UiTM) - Sg Buloh, Bandar Puncak Alam, Selangor
- Erasmus MC, Rotterdam, Netherlands
- Poland (5):
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - UCK, Klinika Pediatrii, Diabetologii i Endokrynologii,, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów
  - SPSK nr 1 im. prof.S.Szyszko w Zabrzu, Zabrze
- South Korea (2):
  - Asan Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and assigned to treatment across 14 sites in 5 countries.
Pre-assignment Details: A total of 47 participants with short stature either born small for gestational age(SGA), Noonan syndrome(NS), Turner syndrome(TS), or idiopathic short stature(ISS) were either treatment naïve or previously treated with growth hormone(GH) were enrolled & exposed to once weekly dosing of somapacitan 0.24 milligrams per kilogram per week(mg/kg/week).
  26-week main phase is followed by 130-week extension phase I. Study was ongoing at data cut-off date(24Nov2024).
Groups:
- SGA_somapacitan (GH Treatment Naïve): Participants with small for gestational age who were treatment naïve subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- SGA_somapacitan (Previously Treated With GH): Participants with small for gestational age who were previously treated with GH, subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- TS_somapacitan (GH Treatment Naïve): Participants with Turner syndrome who were treatment naïve subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- TS_somapacitan (Previously Treated With GH): Participants with Turner syndrome who were previously treated with GH, subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- NS_somapacitan (GH Treatment Naïve): Participants with Noonan syndrome who were treatment naïve subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- NS_somapacitan (Previously Treated With GH): Participants with Noonan syndrome who were previously treated with GH, subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- ISS_somapacitan (GH Treatment Naïve): Participants with idiopathic short stature who were treatment naïve subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
- ISS_somapacitan (Previously Treated With GH): Participants with idiopathic short stature who were were previously treated with GH, subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
Period: Main Trial Period: Weeks 0 to 26
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH) | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH) | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH) | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Started | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9
Full Analysis Set (FAS) | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9
Safety Analysis Set (SAS) | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9
Completed | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension I Period: Weeks 39 Upto 156
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH) | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH) | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH) | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Started | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9
Not completed — Study is ongoing, data is reported till data cut-off 24 Nov 2024 | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants assigned to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH) | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH) | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH) | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH) | Total
Number analyzed (Participants) | 4 | 8 | 3 | 8 | 6 | 7 | 2 | 9 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.50 (2.08) | 11.75 (1.67) | 10.67 (1.15) | 11.00 (1.20) | 12.67 (2.07) | 12.29 (1.50) | 14.50 (0.71) | 11.44 (1.24) | 11.87 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8 | 2 | 2 | 0 | 6 | 26
  Male | 2 | 5 | 0 | 0 | 4 | 5 | 2 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 8 | 3 | 6 | 6 | 7 | 2 | 9 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 7 | 2 | 7 | 5 | 6 | 1 | 6 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs) Reported in Children Born Small for Gestational Age- Weeks 0 to 26
Description: This outcome measure reported number of AEs in children with short stature for indication SGA. Children with SGA are born small for gestational age with insufficient catch-up growth by 2 years of age or older. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
Events | 4 | 10

2. Primary Outcome: Number of Adverse Events Reported for Turner Syndrome (TS)- Weeks 0 to 26
Description: This outcome measure reported number of AEs in participants with short stature for indication TS. TS is a chromosomal disorder which leads to short stature. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
Events | 4 | 18

3. Primary Outcome: Number of Adverse Events Reported for Noonan Syndrome- Weeks 0 to 26
Description: This outcome measure reported number of AEs in participants with short stature for indication NS which is a genetically heterogeneous developmental disorder characterized by postnatally reduced growth and other major disorders. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
Events | 13 | 11

4. Primary Outcome: Number of Adverse Events Reported for Idiopathic Short Stature (ISS)- Weeks 0 to 26
Description: This outcome measure reported number of AEs in participants with short stature for indication ISS. ISS describes short children with normal GH secretion. ISS is a condition in which the height of the individual is more than 2 standard deviations below the corresponding mean height for a given age, sex and population, without evidence of systemic, endocrine, nutritional or chromosomal abnormalities. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
Events | 9 | 22

5. Secondary Outcome: Number of Adverse Events Possibly or Probably Related to Somapacitan Reported for Children Born Small for Gestational Age
Description: This outcome measure reported number of AEs possibly or probably related to somapacitan reported in children with short stature for indication SGA. Children with SGA are born small for gestational age with insufficient catch-up growth by 2 years of age or older. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
Events | 1 | 1

6. Secondary Outcome: Number of Adverse Events Possibly or Probably Related to Somapacitan Reported for Turner Syndrome
Description: This outcome measure reported number of AEs possibly or probably related to somapacitan reported in participants with short stature for indication TS. TS is a chromosomal disorder which leads to short stature. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
Events | 0 | 0

7. Secondary Outcome: Number of Adverse Events Possibly or Probably Related to Somapacitan Reported for Noonan Syndrome
Description: This outcome measure reported number of AEs possibly or probably related to somapacitan reported in participants with short stature for indication NS. An NS is a genetically heterogeneous developmental disorder characterized by postnatally reduced growth and other major disorders. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
Events | 3 | 2

8. Secondary Outcome: Number of Adverse Events Possibly or Probably Related to Somapacitan Reported for Idiopathic Short Stature
Description: This outcome measure reported number of AEs possibly or probably related to somapacitan in participants with short stature for indication ISS. ISS describes short children with normal GH secretion and it is a condition in which the height of the individual is more than 2 standard deviations below the corresponding mean height for a given age, sex and population, without evidence of systemic, endocrine, nutritional or chromosomal abnormalities. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 26
Population: Safety analysis set included all participants who were exposed to study treatment.
Measure: Number; unit: Events
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
Events | 0 | 1

9. Secondary Outcome: Number of Adverse Events Reported Long-term Safety for Children Born Small for Gestational Age- Weeks 0 to 156
Description: This outcome measure reported long-term safety in terms of number of AEs in children with short stature for indication SGA. Children with SGA are born small for gestational age with insufficient catch-up growth by 2 years of age or older. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 156
Reporting Status: Not Posted, anticipated posting 2027-12

10. Secondary Outcome: Number of Adverse Events Reported Long-term Safety for Turner Syndrome- Weeks 0 to 156
Description: This outcome measure reported long-term safety in terms of number of AEs in participants with short stature for indication TS. TS is a chromosomal disorder which leads to short stature. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 156
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: Number of Adverse Events Reported Long-term Safety for Noonan Syndrome- Weeks 0 to 156
Description: This outcome measure reported long-term safety in terms of number of AEs in participants with short stature for indication NS which is a genetically heterogeneous developmental disorder characterized by postnatally reduced growth and other major disorders. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 156
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: Number of Adverse Events Reported Long-term Safety for Idiopathic Short Stature- Weeks 0 to 156
Description: This outcome measure reported long-term safety in terms of number of AEs in participants with short stature for indication ISS. ISS describes short children with normal GH secretion. ISS is a condition in which the height of the individual is more than 2 standard deviations below the corresponding mean height for a given age, sex and population, without evidence of systemic, endocrine, nutritional or chromosomal abnormalities. An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment.
Time Frame: From baseline (Week 0) to Week 156
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Height Velocity Reported Children Born Small for Gestational Age
Description: This outcome measure reported height velocity in children with short stature for indication SGA. Height velocity at week 26 was derived as: (height at 26 weeks visit - height at baseline)/ (time from baseline to 26 weeks visit in years).
Time Frame: From Baseline (Week 0) to Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: centimeters per year (cm/year)
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
centimeters per year (cm/year) | 11.3 (3.8) | 9.5 (2.0)

14. Secondary Outcome: Height Velocity Reported for Turner Syndrome
Description: This outcome measure reported height velocity in children with short stature for indication TS. Height velocity at week 26 was derived as: (height at 26 weeks visit - height at baseline)/ (time from baseline to 26 weeks visit in years).
Time Frame: From Baseline (Week 0) to Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
cm/year | 10.2 (2.2) | 5.8 (2.0)

15. Secondary Outcome: Height Velocity Reported for Noonan Syndrome
Description: This outcome measure reported height velocity in children with short stature for indication NS. Height velocity at week 26 was derived as: (height at 26 weeks visit - height at baseline)/(time from baseline to 26 weeks visit in years).
Time Frame: From Baseline (Week 0) to Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
cm/year | 9.1 (2.3) | 6.4 (2.0)

16. Secondary Outcome: Height Velocity Reported for Idiopathic Short Stature
Description: This outcome measure reported height velocity in children with short stature for indication ISS. Height velocity at week 26 was derived as: (height at 26 weeks visit - height at baseline)/ (time from baseline to 26 weeks visit in years).
Time Frame: From Baseline (Week 0) to Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
cm/year | 9.2 (3.5) | 7.9 (2.4)

17. Secondary Outcome: Change in Height Standard Deviation Scores (SDS) Reported for Children Born Small for Gestational Age
Description: This outcome measure reported height standard deviation scores in children with short stature for indication SGA. Height SDS at Week 26 was derived as the Height SDS value at baseline (Week 0) subtracted from the Height SDS value at Week 26. Height SDS is derived as: Height SDSi = ({[Heighti/population median]^Skewness}-1)/(Skewness∗population SD); where i indicates the visit and SD indicates the standard deviation (SD). The population median and standard deviation are the ones corresponding to the age at visit i. The population median and standard deviation and skewness are based on reference data. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height. The positive score indicates that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
standard deviation score | 0.50 (0.21) | 0.24 (0.13)

18. Secondary Outcome: Change in Height Standard Deviation Scores Reported for Turner Syndrome
Description: This outcome measure reported height standard deviation scores in children with short stature for indication TS. Height SDS at Week 26 was derived as the Height SDS value at baseline (Week 0) subtracted from the Height SDS value at Week 26. Height SDS is derived as: Height SDSi = ({[Heighti/population median]^Skewness}-1)/(Skewness∗population SD); where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The population median and standard deviation and skewness are based on reference data. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height. The positive score indicates that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
standard deviation score | 0.40 (0.30) | 0.00 (0.23)

19. Secondary Outcome: Change in Height Standard Deviation Scores Reported for Noonan Syndrome
Description: This outcome measure reported height standard deviation scores in children with short stature for indication NS. Height SDS at Week 26 was derived as the Height SDS value at baseline (Week 0) subtracted from the Height SDS value at Week 26. Height SDS is derived as: Height SDSi = ({[Heighti/population median]^Skewness}-1)/(Skewness∗population SD); where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The population median and standard deviation and skewness are based on reference data. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height. The positive score indicates that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
standard deviation score | 0.35 (0.26) | 0.11 (0.14)

20. Secondary Outcome: Change in Height Standard Deviation Scores Reported for Idiopathic Short Stature
Description: This outcome measure reported height standard deviation scores in children with short stature for indication ISS. Height SDS at Week 26 was derived as the Height SDS value at baseline (Week 0) subtracted from the Height SDS value at Week 26. Height SDS is derived as: Height SDSi = ({[Heighti/population median]^Skewness}-1)/(Skewness∗population SD); where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The population median and standard deviation and skewness are based on reference data. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height. The positive score indicates that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
standard deviation score | 0.22 (0.15) | 0.14 (0.18)

21. Secondary Outcome: Change in Height Velocity Standard Deviation Scores Reported Separately for Children Born Small for Gestational Age
Description: This outcome measure reported change in height velocity SDS in children with short stature for indication SGA. Change in height velocity SDS at week 26 was calculated as the height velocity SDS value at baseline Week 0 subtracted from the height velocity SDS value at Week 26. Height Velocity SDS is derived as: HV SDSi = (HVi - population mean HV)/population SD; where i indicates the visit. The population mean and standard deviation corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height velocity. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
standard deviation score | 3.53 (2.49) | 1.04 (1.18)

22. Secondary Outcome: Change in Height Velocity Standard Deviation Scores Reported Separately for Turner Syndrome
Description: This outcome measure reported change in height velocity SDS in children with short stature for indication TS. Change in height velocity SDS at week 26 was calculated as the height velocity SDS value at baseline (Week 0) subtracted from the height velocity SDS value at Week 26. Height Velocity SDS is derived as: HV SDSi = (HVi - population mean HV)/population SD; where i indicates the visit. The population mean and standard deviation corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height velocity. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Groups:
- TS_somapacitan (GH Treatment Naïve): TS_somapacitan (GH Treatment Naïve) Participants with Turner syndrome who were treatment naïve subcutaneously received a dose of 0.24 mg/kg/week somapacitan once weekly for 26-week main phase followed by an ongoing 130-week extension phase I.
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
standard deviation score | 3.45 (1.41) | -0.48 (1.84)

23. Secondary Outcome: Change in Height Velocity Standard Deviation Scores Reported for Noonan Syndrome
Description: This outcome measure reported change in height velocity SDS in children with short stature for indication NS. Change in height velocity SDS at Week 26 was the Height Velocity SDS value at baseline (Week 0) subtracted from the Height Velocity SDS value at Week 26. Height Velocity SDS is derived as: HV SDSi = (HVi - population mean HV)/population SD; where i indicates the visit. The population mean and standard deviation corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height velocity. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
standard deviation score | 3.43 (2.75) | 0.22 (0.93)

24. Secondary Outcome: Change in Height Velocity Standard Deviation Scores Reported Separately for Idiopathic Short Stature
Description: This outcome measure reported change in height velocity SDS in children with short stature for indication ISS. Change in height velocity SDS at Week 26 was the Height Velocity SDS value at baseline (Week 0) subtracted from the Height Velocity SDS value at Week 26. Height Velocity SDS is derived as: HV SDSi = (HVi - population mean HV)/population SD; where i indicates the visit. The population mean and standard deviation corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater height velocity. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
standard deviation score | 2.89 (0.85) | -0.32 (1.90)

25. Secondary Outcome: Change in Insulin-like Growth Factor 1 (IGF-1) Standard Deviation Score Reported for Children Born Small for Gestational Age
Description: This outcome measure reported change in IGF-1 SDS in children with short stature for indication SGA. Change in IGF-I SDS was derived as IGF-1 SDS value at baseline Week 0 subtracted from the IGF-I SDS value at Week 26. IGF-I SDS is derived as: IGF - I SDSi = ({[IGF - I i]/population median}^Skewness - 1)/ Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGF-1. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
standard deviation score | 1.61 (1.52) | 1.39 (1.14)

26. Secondary Outcome: Change in Insulin-like Growth Factor 1 Standard Deviation Score Reported for Turner Syndrome
Description: This outcome measure reported change in IGF-1 SDS in children with short stature for indication TS. Change in IGF-I SDS was derived as IGF-1 SDS value at baseline Week 0 subtracted from the IGF-I SDS value at Week 26. IGF-I SDS is derived as: IGF - I SDSi = ({[IGF - I i]/population median}^Skewness - 1)/ Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGF-1. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
standard deviation score | 0.88 (0.43) | -0.09 (1.52)

27. Secondary Outcome: Change in Insulin-like Growth Factor 1 Standard Deviation Score Reported for Noonan Syndrome
Description: This outcome measure reported change in IGF-1 SDS in children with short stature for indication NS. Change in IGF-I SDS was derived as IGF-1 SDS value at baseline Week 0 subtracted from the IGF-I SDS value at Week 26. IGF-I SDS is derived as: IGF - I SDSi = ({[IGF - I i]/population median}^Skewness - 1)/ Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGF-1. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
standard deviation score | 1.01 (1.38) | 2.23 (1.87)

28. Secondary Outcome: Change in Insulin-like Growth Factor 1 Standard Deviation Score Reported Separately for Idiopathic Short Stature
Description: This outcome measure reported change in IGF-1 SDS in children with short stature for indication ISS. Change in IGF-I SDS was derived as IGF-1 SDS value at baseline Week 0 subtracted from the IGF-I SDS value at Week 26. IGF-I SDS is derived as: IGF - I SDSi = ({[IGF - I i]/population median}^Skewness - 1)/ Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGF-1. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
standard deviation score | 2.79 (0.52) | 1.66 (1.28)

29. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein-3 (IGFBP-3) SDS Reported for Children Born Small for Gestational Age
Description: This outcome measure reported change in IGFBP-3 scores in children with short stature for indication SGA. Change in IGFBP-3 SCS at Week 26 was derived as the IGFBP-3 SDS value at baseline Week 0 subtracted from IGFBP-3 SDS value at Week 26. IGFBP-3 SDS is derived as: IGFBP - 3 SDSi = ({[IGFBP - 3 i/population median]^Skewness} - 1)/Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGFBP-3. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
standard deviation score | 0.69 (0.93) | 1.22 (1.00)

30. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein-3 SDS Reported for Turner Syndrome
Description: This outcome measure reported change in IGFBP-3 scores in children with short stature for indication TS. Change in IGFBP-3 SCS at Week 26 was derived as the IGFBP-3 SDS value at baseline Week 0 subtracted from IGFBP-3 SDS value at Week 26. IGFBP-3 SDS is derived as: IGFBP - 3 SDSi = ({[IGFBP - 3 i/population median]^Skewness} - 1)/Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGFBP-3. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention. Here 'Number of participants analysed' signifies number of participants with available data for particular timepoint.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 7
standard deviation score | 0.39 (0.48) | 0.05 (1.45)

31. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein-3 SDS Reported for Noonan Syndrome
Description: This outcome measure reported change in IGFBP-3 scores in children with short stature for indication NS. Change in IGFBP-3 SCS at Week 26 was derived as the IGFBP-3 SDS value at baseline Week 0 subtracted from IGFBP-3 SDS value at Week 26. IGFBP-3 SDS is derived as: IGFBP - 3 SDSi = ({[IGFBP - 3 i/population median]^Skewness} - 1)/Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGFBP-3. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
standard deviation score | 0.66 (0.97) | 0.67 (1.08)

32. Secondary Outcome: Change in Insulin-like Growth Factor Binding Protein-3 SDS Reported for Idiopathic Short Stature
Description: This outcome measure reported change in IGFBP-3 scores in children with short stature for indication ISS. Change in IGFBP-3 SCS at Week 26 was derived as the IGFBP-3 SDS value at baseline Week 0 subtracted from IGFBP-3 SDS value at Week 26. IGFBP-3 SDS is derived as: IGFBP - 3 SDSi = ({[IGFBP - 3 i/population median]^Skewness} - 1)/Skewness ∗ population SD; where i indicates the visit. The population median and standard deviation are the ones corresponding to the age at visit i. The score ranges from -10 (minimum) to +10 (maximum), where the greater value indicated greater IGFBP-3. The positive score indicated that the value is closer to or above the reference population compared to baseline.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
standard deviation score | 1.22 (0.18) | 1.08 (1.43)

33. Secondary Outcome: Weekly Average Somapacitan Concentration (Cavg) Reported for Children Born Small for Gestational Age
Description: The steady state pharmacokinetics in terms of Cavg was evaluated for once-weekly somapacitan in children born small for gestational age who were either naïve or non-naïve to GH treatment.
Time Frame: Weeks 4, 8, 13, 20 and 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 4 | 8
nanograms per milliliter (ng/mL)
  Week 4 | 518.948 (58.993) | 339.226 (205.265)
  Week 8 | 1.800 (0.857) | 2.204 (0.556)
  Week 13 | 62.280 (92.161) | 78.530 (79.022)
  Week 20 | 2.345 (1.331) | 4.123 (3.263)
  Week 26 | 5.928 (4.904) | 8.364 (5.075)

34. Secondary Outcome: Weekly Average Somapacitan Concentration (Cavg) Reported for Turner Syndrome
Description: The steady state pharmacokinetics in terms of Cavg was evaluated for once-weekly somapacitan in children with Turner Syndrome who were either naïve or non-naïve to GH treatment.
Time Frame: Weeks 4, 8, 13, 20 and 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 3 | 8
nanograms per milliliter (ng/mL)
  Week 4 | 287.777 (191.086) | 384.130 (252.372)
  Week 8 | 2.187 (0.335) | 3.285 (2.018)
  Week 13 | 75.400 (125.123) | 93.753 (162.274)
  Week 20 | 2.487 (1.232) | 2.871 (1.018)
  Week 26 | 4.363 (2.890) | 8.574 (5.304)

35. Secondary Outcome: Weekly Average Somapacitan Concentration (Cavg) Reported for Noonan Syndrome
Description: The steady state pharmacokinetics in terms of Cavg was evaluated for once-weekly somapacitan in children with Noonan Syndrome who were either naïve or non-naïve to GH treatment.
Time Frame: Weeks 4, 8, 13, 20 and 26
Population: Full analysis set included all participants assigned to study intervention.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 6 | 7
nanograms per milliliter (ng/mL)
  Week 4 | 249.278 (225.237) | 254.626 (175.518)
  Week 8 | 3.102 (2.197) | 31.343 (58.845)
  Week 13 | 102.647 (164.113) | 134.501 (188.934)
  Week 20 | 34.043 (69.759) | 3.869 (2.376)
  Week 26 | 13.057 (22.222) | 42.834 (58.984)

36. Secondary Outcome: Weekly Average Somapacitan Concentration (Cavg) Reported for Idiopathic Short Stature
Description: The steady state pharmacokinetics in terms of Cavg was evaluated for once-weekly somapacitan in children with idiopathic short stature who were either naïve or non-naïve to GH treatment.
Time Frame: Weeks 4, 8, 13, 20 and 26
Population: Full analysis set included all participants assigned to study intervention. Here, 'Number Analyzed' signifies number of participants with available data for particular timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
Number analyzed (Participants) | 2 | 9
nanograms per milliliter (ng/mL)
  Week 4 | 344.415 (313.128) | 401.444 (178.512)
  Week 8 | 9.535 (0.940) | 57.152 (145.426)
  Week 13 | 403.525 (156.235) | 74.361 (65.211)
  Week 20 | 7.070 (3.564) | 4.876 (4.495)
  Week 26: number analyzed (Participants) | 1 | 9
  Week 26 | 16.630 (NA) — Since only a single participant was assessed in this arm, the standard deviation could not be calculated and is reported as 'Not Applicable'. | 16.461 (15.509)

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) up to Week 94 (approximately, Data cut off date: 24Nov2024)
Description: An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study drug, whether or not considered related to the study treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of an study treatment. Safety analysis set included all participants who were exposed to study treatment.
Arm/Group | SGA_somapacitan (GH Treatment Naïve) | SGA_somapacitan (Previously Treated With GH) | TS_somapacitan (GH Treatment Naïve) | TS_somapacitan (Previously Treated With GH) | NS_somapacitan (GH Treatment Naïve) | NS_somapacitan (Previously Treated With GH) | ISS_somapacitan (GH Treatment Naïve) | ISS_somapacitan (Previously Treated With GH)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/3 | 0/8 | 0/6 | 0/7 | 0/2 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/8 | 0/3 | 1/8 | 0/6 | 0/7 | 0/2 | 1/9
Other Adverse Events (participants affected / at risk) | 3/4 | 5/8 | 2/3 | 7/8 | 4/6 | 6/7 | 2/2 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SGA_somapacitan (GH Treatment Naïve) (N=4) | SGA_somapacitan (Previously Treated With GH) (N=8) | TS_somapacitan (GH Treatment Naïve) (N=3) | TS_somapacitan (Previously Treated With GH) (N=8) | NS_somapacitan (GH Treatment Naïve) (N=6) | NS_somapacitan (Previously Treated With GH) (N=7) | ISS_somapacitan (GH Treatment Naïve) (N=2) | ISS_somapacitan (Previously Treated With GH) (N=9)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal microorganism overgrowth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SGA_somapacitan (GH Treatment Naïve) (N=4) | SGA_somapacitan (Previously Treated With GH) (N=8) | TS_somapacitan (GH Treatment Naïve) (N=3) | TS_somapacitan (Previously Treated With GH) (N=8) | NS_somapacitan (GH Treatment Naïve) (N=6) | NS_somapacitan (Previously Treated With GH) (N=7) | ISS_somapacitan (GH Treatment Naïve) (N=2) | ISS_somapacitan (Previously Treated With GH) (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Accidental underdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (14)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac imaging procedure abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema infectiosum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insulin-like growth factor increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intellectual disability (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Precocious puberty (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Product administration error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 2 (3)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT05723835/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT05723835/SAP_001.pdf